CLINICAL TRIAL: NCT05860114
Title: An Open-label, Single-center, Study in Healthy Subjects to Evaluate the Plasma and Urine Pharmacokinetics of Givinostat and Its Metabolites Following Single and Multiple Oral Doses of Givinostat (Part 3).
Brief Title: Givinostat and Metabolites Pharmacokinetics in Urine and Plasma (Part 3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITF/2357/55 - PART 3; 2021-005756-11 (EudraCT Number)
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-07

CONDITIONS: Drug Drug Interaction
Keywords: PK; Pharmacokinetics; Givinostat; Givinostat metabolites
MeSH Terms: interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Masking Description: The study was conducted as open label. Blinding procedures were not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Givinostat (single-dose and multiple-dose) (Experimental): On Days 1 and 13, Givinostat 50 mg as oral suspension was administered as a single dose, in the morning. On Days 5-12 Givinostat 50 mg as oral suspension was administered twice-daily, in the morning and in the evening, as a multiple dose.
  PK parameters values following:
  * single oral dose administration of Givinostat (Day 1) and
  * multiple oral dose administration of Givinostat (Day 5 to Day 12, with values reported at Day 13) were assessed and reported.
  Interventions: Drug: Givinostat

INTERVENTIONS:
Drug: Givinostat — Drug: ITF2357 Givinostat 10mg/mL Dose: 10mg/mL; Dosage form: oral suspension
  On days 1 and 13 givinostat was administered in the morning, following an overnight fasting of at least 8 hours and subjects remained fasted until at least 4 hours post-dose. Moreover the subjects were in a semi-recumbent position and remained semi-recumbent until at least 4 hours post-dose.No fluids were allowed from 1 hour before dosing until 2 hours post-dose. Water was provided ad libitum at all other times.
  From Day 5 to Day 12, subjects received givinostat 50 mg as oral suspension, twice a day, in the morning and in the evening.
  Other Names: ITF2357

SUMMARY:
Primary objective:

To evaluate the plasma and urine PK of Givinostat following multiple oral doses of Givinostat.

Secondary objective:

To assess the safety and tolerability multiple oral doses of Givinostat.

DETAILED DESCRIPTION:
This study was planned as a phase I, open-label, 3-part, fixed-sequence, nonrandomized study in healthy male and female subjects. The study (Part 3) aimed at assessing Givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) plasma and urine concentrations and thereof derived pharmacokinetic parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Day 5 to Day 12, with measures reported at Day 13, before single-dose administration). More precisely, Gmean and corresponding 95% CI of Givinostat plasma and urine concentration and Givinostat metabolites plasma concentration versus time profiles following single (Day 1) and multiple-dose (Day 5 to Day 12, with measures reported at Day 13) administration of Givinostat are reported using Linear Scale and Semi-Logarithmic Scale.

Descriptive statistics of Givinostat plasma pharmacokinetic parameters and Givinostat metabolites PK parameters following single-dose administration of Givinostat (Day 1) and following multiple-dose administration of Givinostat (Days 5-12, with measures reported at Day 13) were calculated.

Descriptive statistics of Givinostat and its metabolites urinary excretion profile following single-dose administration of Givinostat (Day 1) and following multiple dose administration of Givinostat (Days 5-12, with measures reported at Day 13) were calculated.

Descriptive statistics of Givinostat and its metabolites cumulative amount of urinary excretion profile following single-dose administration of Givinostat (Day 1) and following multiple-dose administration of Givinostat (Days 5-12, with measures reported at Day 13) were also calculated using linear scales.

ELIGIBILITY:
Inclusion Criteria:

* A subject was considered eligible for the study if he/she fulfilled all the inclusion criteria:

  1. Subject's written informed consent obtained prior to any study-related procedure.
  2. Male or female subject, ≥18 and ≤55 years of age, at the time of signing the informed consent.
  3. Body mass index (BMI) of 18.5 to 32.0 kg/m2 inclusive, and body weight ≥55 kg and ≤100 kg for females and body weight ≥60 kg and ≤110 kg for males.
  4. Non-smoker or ex-smoker (i.e. someone who abstained from using tobaccoor nicotine-containing products for at least 3 months prior to Screening).
  5. No clinically relevant diseases.
  6. No major surgery within 4 weeks prior to dosing.
  7. No clinically relevant abnormalities on physical examination.
  8. No clinically relevant abnormalities on 12-lead ECG.
  9. No clinically relevant abnormalities on clinical laboratory tests.
  10. Negative test results for anti-Human Immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), Hepatitis B surface antigen (HBsAg) and anti-Hepatitis C virus antibodies (anti-HCVAb).
  11. Female subjects are eligible if they are of non-childbearing potential or agree to use a non-hormonal highly effective contraceptive method from 28 days prior to Screening until at least 90 days after the last study drug administration. Nonchildbearing potential female is defined as:

      1. Menopausal, i.e. no menses for ≥ 12 months without an alternative medical cause other than menopause, and a high FSH level.
      2. Pre-menopausal female with documented hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy.

      A non-hormonal effective contraceptive method is defined as:
      1. Intrauterine device.
      2. Bilateral tubal occlusion.
      3. Total abstinence of heterosexual intercourse, in accordance with the lifestyle of the subject.
      4. Vasectomized partner, who has received medical assessment of the surgical success, or clinically diagnosed infertile partner.
  12. Male subjects who are sexually active with a female partner of childbearing potential (pregnant or non-pregnant) must use contraception (condom) from investigational product administration up to at least 90 days following the last study drug administration.
  13. Male subjects must ensure that his non-pregnant female partner of childbearing potential agrees to consistently and correctly use for the same period a highly effective method of contraception.
  14. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
  15. Willingness and capability to comply with the requirements of the study and ability to understand the study procedures and the risks involved.

Exclusion Criteria:

A subject was excluded from the study if he/she fulfilled any of the exclusion criteria:

At Screening

1. Previous use of givinostat.
2. History of anaphylaxis reaction or clinically significant drug hypersensitivity reaction (e.g., angioedema, Stevens-Johnson syndrome, acute generalized exanthematous pustulosis, drug-induced hypersensitivity syndrome, druginduced neutropenia).
3. Known history of hypersensitivity and/or allergic reactions to givinostat, histone deacetylases (HDAC) inhibitors or to any excipient in the formulation.
4. History of sorbitol intolerance, sorbitol malabsorption or fructose intolerance.
5. Any medical condition (e.g. gastrointestinal, renal or hepatic, including peptic ulcer, inflammatory bowel disease or pancreatitis) or surgical condition (e.g. cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion) or subject safety.
6. Systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg, or pulse rate lower than 50 or over 100 bpm.
7. QTcF ˃450 msec.
8. Subjects with history of cardiac arrhythmias (documented), family history of sudden cardiac death or history of additional risk factors for torsades-depointes (e.g. heart failure, hypokalemia, long QT syndrome).
9. Having an estimated glomerular filtration (eGFR) < 90 mL/min, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average surface area of 1.73 m2.
10. Any of the following abnormal laboratory test values:

    1. Platelet count below the lower limit of the normal range (LLN)
    2. Total white blood cells count below the LLN
    3. Hemoglobin below the LLN
    4. Triglycerides above the upper limit of normal range (ULN)
    5. Potassium or magnesium below the LLN
11. Positive urine alcohol, drugs-of-abuse or cotinine screen tests.
12. Positive serum pregnancy test.
13. If woman, she is breast-feeding.
14. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (i.e. more than 14 units of alcohol per week for males or more than 7 units for females).
15. History of drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs [such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives] within 1 year prior to screening.
16. Participation in any clinical trial within the previous 2 months.
17. Participation in more than 2 clinical trials within the previous 12 months.
18. Blood donation or significant blood loss (≥ 450 mL) due to any reason or had plasmapheresis within the previous 2 months.
19. Veins unsuitable for intravenous puncture on either arm.
20. Difficulty in swallowing capsules, tablets or suspensions.
21. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

    At Admission to Treatment Period
22. Any clinically relevant abnormalities on clinical laboratory tests.
23. Positive urine alcohol, drugs-of-abuse or cotinine screen tests.
24. Positive urine pregnancy test.
25. Positive or inconclusive SARS-CoV-2 test prior to admission.
26. Use of prescription or non-prescription medicinal products within the previous 28 days or within 5-half-lives of the medicinal product, whichever is longer.
27. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Blueclinical, Ltd.
Locations (1):
- Hospital da Prelada, 3rd Floor & East Wing 4th Floor Rua Sarmento de Beires, Porto, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 subjects were screened for participation. Eight (8) subjects (2 women and 6 men) were admitted to study Part 3.
Groups:
- Givinostat (Single-dose and Multiple-dose): On Day 1 and Day 13, Givinostat 50 mg as oral suspension was administered as a single dose, in the morning.
  On Days 5-12 Givinostat 50 mg as oral suspension was administered twice-daily, in the morning and in the evening, as a multiple dose.
  Givinostat: Drug: ITF2357 Givinostat 10mg/mL Dose: 10mg/mL; Dosage form: oral suspension
Period: Overall Study
Arm/Group | Givinostat (Single-dose and Multiple-dose)
Started | 8
Safety Analysis Population | 8
Single-dose PK Population | 8
Multiple-dose PK Population | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eight (8) subjects were enrolled in Part 3 of the study and provided evaluable pharmacokinetic data for the Givinostat single-dose administration (Day 1) or multiple-dose administration (Day 13), without deviations affecting pharmacokinetic interpretation. They constitute the Part 3 (Single-Dose or multiple-dose) Pharmacokinetic Analysis Population.
Groups:
- Givinostat (Single-dose or Multiple-dose): On day 1, givinostat 50 mg as oral suspension was administered as a single dose, in the morning. On Days 5-12 givinostat 50 mg as oral suspension was administered twice-daily, in the morning and in the evening, as a multiple dose. On day 13 givinostat 50 mg as oral suspension was administered as a single dose, in the morning.
  Givinostat: Drug: ITF2357 Givinostat 10mg/mL Dose: 10mg/mL; Dosage form: oral suspension
Arm/Group | Givinostat (Single-dose or Multiple-dose)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Portugal | 8

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pharmacokinetic (PK) Parameters of Givinostat, Following First Single-dose Administration of Givinostat: Cmax
Description: Cmax is the Maximum Observed Plasma Concentration. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 22 blood samples were collected as follows:
  - 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Days 1, for the determination of Givinostat and its metabolites plasma concentrations using a validated LC-MS/MS analytical method.
  Summary Statistics for the main PK parameters, like Cmax, Following Single-Dose Administration of Givinostat (Day 1) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 1.
Population: Eight (8) subjects were enrolled in Part 3 of the study and provided evaluable pharmacokinetic data for the Givinostat single-dose administration (Day 1), without deviations affecting pharmacokinetic interpretation. They constitute the Part 3 Single-Dose Pharmacokinetic Analysis Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Givinostat: On Day 1 and Day 13, Givinostat 50 mg as oral suspension was administered as a single dose in the morning. From Day 5 to Day 12, Givinostat 50 mg as oral suspension was administered twice a day, in the morning and in the evening.
- ITF2374; ITF2375; ITF2440; ITF2563: Givinostat plasma metabolite
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL | 48.06 (25.8) | 7.34 (45.7) | 132.20 (40.2) | 88.77 (16.4) | 15.38 (13.8)

2. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose Administration of Givinostat: Tmax
Description: Tmax is the Time to Maximum Observed Concentration.The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 22 blood samples were collected as follows:
  - 22 blood samples at predose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Days 1, for the determination of Givinostat and its metabolites plasma concentrations.
  Summary Statistics for the main PK parameters, like tmax, Following Single-Dose Administration of Givinostat (Day 1) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 1.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours | 1.50 [1.00 to 3.50] | 5.50 [5.00 to 12.00] | 3.50 [2.00 to 4.00] | 9.00 [8.00 to 12.00] | 10.00 [8.00 to 12.00]

3. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose and Following Multiple-Dose Administration of Givinostat: Ctrough
Description: Ctrough is the Pre-dose Plasma Concentration. On Day 1 and Day 13, Givinostat 50 mg as oral suspension was administered as a single dose, in the morning, following an overnight fasting of at least 8 hours and subjects remained fasted until at least 4 hours post-dose. From Day 5 to Day 12 Givinostat 50 mg as oral suspension was administered twice daily.
  A total of 48 blood samples were collected:
  * 22 during single-dose treatment (Day 1, at pre-dose and at the timepoints indicated in the timeframe post-dose) and
  * 26 during the multiple dose treatment (Days 5-12 plus single-dose treatment at Day 13). Of these 26 samples: 22 as per Day 1, and 4 before the morning dose of IMP on Days 9, 10, 11 and 12.
  PK plasma parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 1 and on Day 13.
Population: Eight (8) subjects were enrolled in Part 3 of the study and provided evaluable pharmacokinetic data for the Givinostat single-dose administration (Day 1 and Day 13 in the morning), without deviations affecting pharmacokinetic interpretation. They constitute the Part 3 Pharmacokinetic Analysis Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Givinostat: On Day 1 and Day 13, Givinostat 50 mg as oral suspension was administered as a single dose in the morning following an overnight fasting of at least 8 hours and subjects remained fasted until at least 4 hours post-dose.
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL
  single dose (Day 1) | 6.75 (22.3) | 4.14 (42.6) | 28.47 (53.3) | 81.58 (14.9) | 14.75 (11.1)
  multiple dose (Day 13) | 13.16 (28.7) | 10.18 (50.8) | 56.12 (60.6) | 279.96 (15.6) | 50.11 (18.8)

4. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose and Following Multiple-dose Administration of Givinostat: AUC0-inf.
Description: AUC0-inf is the AUC from Time Zero to Infinity. On Day 1 and Day 13, givinostat 50 mg as oral suspension was administered as a single dose, in the morning, following an overnight fasting of at least 8 hours and subjects remained fasted until at least 4 hours post-dose. From Day 5 to Day 12 givinostat 50 mg as oral suspension was administered twice daily.
  A total of 48 blood samples were collected:
  * 22 during single-dose treatment (Day 1, at pre-dose and at the timepoints indicated in the timeframe post-dose) and
  * 26 during the multiple dose treatment (Days 5-12 plus single-dose treatment at Day 13). Of these 26 samples: 22 as per Day 1, and 4 before the morning dose of IMP on Days 9, 10, 11 and 12.
  PK plasma parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: as for outcome 3
Population: Eight (8) subjects were enrolled in Part 3 of the study and provided evaluable pharmacokinetic data for the givinostat single-dose administration (Day 1) and multiple-dose administration (Day 13), without deviations affecting pharmacokinetic interpretation. They constitute the Part 3 Single-Dose and Multiple-Dose Pharmacokinetic Analysis Population, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h*ng/mL
  Single-dose (Day 1) | 305.72 (21.0) | 99.01 (49.1) | 1239.34 (47.8) | 2431.31 (12.1) | 457.95 (13.4)
  Multiple-dose (Day 13) | 562.42 (17.5) | 337.71 (53.2) | 2754.89 (77.8) | 9526.56 (30.2) | 1715.62 (23.0)

5. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose and Following Multiple-dose Administration of Givinostat: AUC0-t.
Description: AUC0-t is the AUC from Time Zero to Last Sampling Time with Quantifiable. On Days 1 and 13, Givinostat 50 mg as oral suspension was administered as a single dose, in the morning, following an overnight fasting of at least 8 h and subjects remained fasted until at least 4 h post-dose. From Day 5 to Day 12 Givinostat 50 mg as oral suspension was administered twice daily.
  48 blood samples were collected in total:
  * 22 during single-dose treatment (Day 1, at pre-dose and at the timepoints indicated in the timeframe post-dose),
  * 26 during the multiple dose treatment (Days 5-12 plus single-dose treatment at Day 13). Of these 26 samples: 22 as per Day 1, and 4 before the morning dose of IMP on Days 9, 10, 11 and 12.
  PK plasma parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: as for outcome 3
Population: Eight (8) subjects were enrolled in Part 3 of the study and provided evaluable pharmacokinetic data for the Givinostat single-dose administration (Day 1 and Day 13) and multiple-dose administration (From Day 5 to Day 12), without deviations affecting pharmacokinetic interpretation. They constitute the Part 3 Single-Dose and Multiple-Dose Pharmacokinetic Analysis Population, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h*ng/mL
  Single-dose (Day 1) | 300.45 (21.3) | 93.30 (51.0) | 1223.60 (47.5) | 2345.60 (12.7) | 439.59 (13.0)
  Multiple-dose (Day 13) | 554.78 (17.5) | 328.36 (53.9) | 2609.03 (68.2) | 9262.28 (27.4) | 1681.26 (21.8)

6. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose Administration of Givinostat: AUC0-τ
Description: AUC0-τ is the area under the plasma concentration versus time curve. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 22 blood samples were collected as follows:
  - 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Days 1, for the determination of Givinostat and its metabolites plasma concentrations.
  Summary Statistics for the main PK parameters, like AUC0-τ, Following Single-Dose Administration of Givinostat (Day 1) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h*ng/mL | 245.73 (23.2) | 52.48 (42.2) | 806.71 (40.6) | 681.56 (25.8) | 99.71 (23.1)

7. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose and Following Multiple-dose Administration of Givinostat: %AUCextrap
Description: Area under the curve (AUC) is used to describe the total exposure to a drug. The total AUC (AUC0-∞) is the area under the curve from time 0 extrapolated to infinite time. %AUCextrap is the Residual Area or Percentage of Extrapolated Part of AUC0-∞.
  On Days 1 and 13, givinostat 50 mg as oral suspension was administered as a single dose, in the morning, following an overnight fasting of at least 8 h and subjects remained fasted until at least 4 h post-dose. From Day 5 to Day 12 Givinostat 50 mg as oral suspension was administered twice daily.
  A total of 48 samples were collected as already described. PK plasma parameters following single oral dose administration of givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-∞
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
percentage of AUC0-∞
  Single-dose (Day 1) | 1.69 (21.7) | 5.39 (39.8) | 0.93 (97.7) | 3.46 (20.9) | 3.96 (16.3)
  Multiple-dose (Day 13) | 1.33 (20.6) | 2.56 (45.2) | 2.13 (220.0) | 1.84 (112.1) | 1.53 (82.8)

8. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose and Following Multiple-dose Administration of Givinostat: λz
Description: λz is the Apparent Terminal Elimination Rate Constant. On Day 1 and Day 13, Givinostat 50 mg as oral suspension was administered as a single dose, in the morning, following an overnight fasting of at least 8 hours and subjects remained fasted until at least 4 hours post-dose. From Day 5 to Day 12 Givinostat 50 mg as oral suspension was administered twice daily.
  A total of 48 blood samples were collected:
  * 22 during single-dose treatment (Day 1, at pre-dose and at the timepoints indicated in the timeframe post-dose) and
  * 26 during the multiple dose treatment (Days 5-12 plus single-dose treatment at Day 13). Of these 26 samples: 22 as per Day 1, and 4 before the morning dose of IMP on Days 9, 10, 11 and 12.
  PK plasma parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
1/hour
  Single-dose (Day 1) | 0.097 (15.6) | 0.094 (33.0) | 0.062 (34.2) | 0.060 (15.2) | 0.055 (27.8)
  Multiple-dose (Day 13) | 0.067 (24.8) | 0.064 (22.5) | 0.037 (71.6) | 0.047 (49.8) | 0.052 (31.5)

9. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose Administration of Givinostat: t1/2
Description: t1/2 is the Apparent Terminal Half-Life. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 22 blood samples were collected as follows:
  - 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Days 1, for the determination of Givinostat and its metabolites plasma concentrations.
  Summary Statistics for the main PK parameters, like t1/2, Following Single-Dose Administration of Givinostat (Day 1) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours | 7.16 (15.7) | 7.40 (32.8) | 11.21 (34.4) | 11.65 (15.4) | 12.57 (27.8)

10. Primary Outcome: Plasma PK Parameters of Givinostat, Following First Single-dose Administration of Givinostat: Vd/F
Description: Vd/F is the Apparent volume of distribution. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 22 blood samples were collected as follows:
  - 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Days 1, for the determination of Givinostat and its metabolites plasma concentrations.
  Summary Statistics for the main PK parameters, like Vd/F, Following Single-Dose Administration of Givinostat (Day 1) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Liters | 1690.43 (21.7) | 0000 (0000) | 0000 (0000) | 0000 (0000) | 0000 (0000)

11. Primary Outcome: Plasma PK Parameters of Givinostat, Following Multiple-dose Administration of Givinostat: Cmax,ss
Description: Cmax,ss is the Maximum Observed Plasma Concentration at steady state. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 26 blood samples were collected as follows:
  * 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Day 13, for the determination of Givinostat and its metabolites plasma concentrations.
  * 4 blood samples before the morning dose of on Days 9, 10, 11 and 12, for the determination of pre-dose plasma concentration of Givinostat and its metabolites.
  Summary Statistics for Cmax,ss, Following Multiple-Dose of Givinostat (Days 5-12 plus single-dose at Day 13, with values calculated at Day 13) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 13.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL | 75.50 (27.0) | 20.52 (38.6) | 217.29 (38.1) | 306.60 (15.2) | 55.37 (20.3)

12. Primary Outcome: Plasma PK Parameters of Givinostat, Following Multiple-dose Administration of Givinostat: Tmax,ss
Description: Tmax,ss is the Time of occurrence of Cmax,ss. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported in this platform).
  A total of 26 blood samples were collected as follows:
  * 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Day 13, for the determination of Givinostat and its metabolites plasma concentrations.
  * 4 blood samples before the morning dose of on Days 9, 10, 11 and 12, for the determination of pre-dose plasma concentration of Givinostat and its metabolites.
  Summary Statistics for Tmax,ss, Following Multiple-Dose of Givinostat (Days 5-12 plus single-dose at Day 13, with values calculated at Day 13) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 13.
Population: Eight (8) subjects were enrolled in Part 3 of the study and provided evaluable pharmacokinetic data for the Givinostat multiple-dose administration (Day 13), without deviations affecting pharmacokinetic interpretation. They constitute the Part 3 Multiple-Dose Pharmacokinetic Analysis Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours | 1.50 [1.50 to 3.00] | 5.50 [5.00 to 6.00] | 3.50 [2.05 to 4.00] | 10.00 [4.00 to 12.00] | 9.00 [6.00 to 10.00]

13. Primary Outcome: Plasma PK Parameters of Givinostat, Following Multiple-dose Administration of Givinostat: AUC0-τ,ss
Description: AUC0-τ,ss is the AUC during a Dosing Interval at steady state. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 26 blood samples were collected as follows:
  * 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field the administration of Givinostat (post-dose), on Day 13, for the determination of Givinostat and its metabolites plasma concentrations.
  * 4 blood samples before the morning dose of on Days 9, 10, 11 and 12, for the determination of pre-dose plasma concentration of Givinostat and its metabolites.
  Summary Statistics for AUC0-τ,ss, Following Multiple-Dose of Givinostat (Days 5-12 plus single-dose at Day 13, with values calculated at Day 13) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 13.
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h*ng/mL | 408.55 (16.2) | 179.63 (41.9) | 1518.21 (50.5) | 3395.41 (15.8) | 586.72 (19.3)

14. Primary Outcome: Plasma PK Parameters of Givinostat, Following Multiple-dose Administration of Givinostat: CLss/F.
Description: CLss/F is the Apparent total body clearance at steady state. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  A total of 26 blood samples were collected as follows:
  * 22 blood samples at pre-dose and at the timepoints indicated in the timeframe field after the administration of Givinostat (post-dose), on Day 13, for the determination of Givinostat and its metabolites plasma concentrations.
  * 4 blood samples before the morning dose of on Days 9, 10, 11 and 12, for the determination of pre-dose plasma concentration of Givinostat and its metabolites.
  Summary Statistics for CLss/F, Following Multiple-Dose of Givinostat (Day 13) are reported.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours post dose on Day 13.
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
L/h | 122.38 (16.2) | 0000 (0000) | 0000 (0000) | 00000 (00000) | 00000 (00000)

15. Primary Outcome: Urinary PK Parameters of Givinostat Following First Single-dose and Following Multiple-dose of Givinostat: Rmax.
Description: Rmax is the Maximum urinary excretion rate. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  Urine was collected, beside on Day -1 (baseline), in the following intervals, on Days 1 and 13, for the determination of the amounts of Givinostat and its metabolites excreted in urine: 0h-12h, 12h-24h, 24h-36h, 36h-48h, 48h-72h and 72h-96h post-dose.
  Givinostat and its metabolites urine levels were measured using a validated LC-MS/MS analytical method.
  PK urine parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 hours post-dose on days 1 and 13.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/h
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mg/h
  single-dose (Day 1) | 0.051 (50.8) | 0.015 (25.9) | 0.006 (44.6) | 0.276 (25.9) | 0.107 (23.6)
  multiple-dose (Day 13) | 0.059 (39.8) | 0.043 (30.6) | 0.009 (83.0) | 0.692 (23.7) | 0.319 (28.3)

16. Primary Outcome: Urinary PK Parameters of Givinostat Following First Single-dose and Following Multiple-dose of Givinostat: Tumax
Description: tumax is the Time to Rmax. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  Urine was collected, beside on Day -1 (baseline), in the following intervals, on Days 1 and 13, for the determination of the amounts of Givinostat and its metabolites excreted in urine: 0h-12h, 12h-24h, 24h-36h, 36h-48h, 48h-72h and 72h-96h post-dose.
  Givinostat and its metabolites urine levels were measured using a validated LC-MS/MS analytical method.
  PK urine parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 hours post-dose on days 1 and 13.
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours
  single-dose (Day 1) | 6.00 [6.00 to 6.00] | 6.00 [6.00 to 18.00] | 6.00 [6.00 to 6.00] | 6.00 [6.00 to 18.00] | 12.00 [6.00 to 18.00]
  multiple-dose (Day 13) | 6.00 [6.00 to 6.00] | 6.00 [6.00 to 6.00] | 6.00 [6.00 to 6.00] | 12.00 [6.00 to 18.00] | 18.00 [6.00 to 18.00]

17. Primary Outcome: Urinary PK Parameters of Givinostat Following First Single-dose and Following Multiple-dose of Givinostat: AmtCUM
Description: AmtCUM is the Cumulative amount of drug excreted in urine. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  Urine was collected, beside on Day -1 (baseline), in the following intervals, on Days 1 and 13, for the determination of the amounts of Givinostat and its metabolites excreted in urine: 0h-12h, 12h-24h, 24h-36h, 36h-48h, 48h-72h and 72h-96h post-dose.
  Givinostat and its metabolites urine levels were measured using a validated LC-MS/MS analytical method.
  PK urine parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 hours post-dose on days 1 and 13.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mg
  single-dose (Day 1) | 0.782 (39.2) | 0.417 (24.9) | 0.093 (49.6) | 9.179 (15.6) | 3.985 (18.6)
  multiple-dose (Day 13) | 1.037 (32.6) | 1.201 (39.8) | 0.184 (85.9) | 26.627 (20.2) | 12.208 (18.3)

18. Primary Outcome: Urinary PK Parameters of Givinostat Following First Single-dose and Following Multiple-dose of Givinostat: AURC0-t
Description: AURC0-t is the Area under the urine excretion curve from time zero to last measurable observed excretion rate. The unit of measure is mg because the value measured is an amount. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  Urine was collected, beside on Day -1 (baseline), in the following intervals, on Days 1 and 13, for the determination of the amounts of Givinostat and its metabolites excreted in urine: 0h-12h, 12h-24h, 24h-36h, 36h-48h, 48h-72h and 72h-96h post-dose.
  Givinostat and its metabolites urine levels were measured using a validated LC-MS/MS analytical method.
  PK urine parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 hours post-dose on days 1 and 13.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mg
  single-dose (Day 1) | 0.532 (31.1) | 0.354 (27.4) | 0.063 (55.3) | 8.019 (16.6) | 3.571 (19.9)
  multiple-dose (Day 13) | 0.773 (30.6) | 1.027 (41.1) | 0.142 (89.0) | 23.836 (19.6) | 10.961 (18.2)

19. Primary Outcome: Urinary PK Parameters of Givinostat Following First Single-dose and Following Multiple-dose of Givinostat: REC%
Description: REC% is the Percentage of drug recovered in urine. The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  Urine was collected, beside on Day -1 (baseline), in the following intervals, on Days 1 and 13, for the determination of the amounts of Givinostat and its metabolites excreted in urine: 0h-12h, 12h-24h, 24h-36h, 36h-48h, 48h-72h and 72h-96h post-dose.
  Givinostat and its metabolites urine levels were measured using a validated LC-MS/MS analytical method.
  PK urine parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 hours post-dose on days 1 and 13.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Percentage of drug
  single-dose (Day 1) | 1.565 (39.1) | 0.868 (24.9) | 0.193 (49.8) | 30.072 (15.6) | 18.852 (18.6)
  multiple-dose (Day 13) | 2.073 (32.6) | 2.496 (39.8) | 0.380 (86.3) | 87.228 (20.2) | 57.755 (18.3)

20. Primary Outcome: Urinary PK Parameters of Givinostat Following First Single-dose and Following Multiple-dose of Givinostat: CLr/F
Description: The Givinostat metabolites were: ITF2374, ITF2375, ITF2440, ITF2563 (not reported on this platform).
  Urine was collected, beside on Day -1 (baseline), in the following intervals, on Days 1 and 13, for the determination of the amounts of Givinostat and its metabolites excreted in urine: 0h-12h, 12h-24h, 24h-36h, 36h-48h, 48h-72h and 72h-96h post-dose.
  Givinostat and its metabolites urine levels were measured using a validated LC-MS/MS analytical method. PK urine parameters following single oral dose administration of Givinostat (Day 1) and following multiple oral dose administration of Givinostat (Days 5-12 plus single-dose treatment at Day 13, with values on multiple-dose treatment reported at Day 13) were assessed.
Time Frame: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 hours post-dose on days 1 and 13.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
L/h
  single-dose (Day 1) | 2.604 (28.6) | 4.473 (44.1) | 0.076 (26.8) | 3.913 (23.7) | 9.065 (25.8)
  multiple-dose (Day 13) | 1.868 (25.4) | 3.656 (26.5) | 0.070 (20.0) | 2.875 (18.3) | 7.261 (17.0)

21. Secondary Outcome: Incidence and Severity of Treatment Emergent Adverse Events
Description: An AE was considered as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily imply a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The period of observation for the collection of medical occurrences extended from the time when the subject gave Informed Consent until the follow-up visit.
Time Frame: Throughout the study, until 10-14 days after EoS (Day 17), i.e. till Days 27-31
Population: The Safety (SAF) population consisted of all randomized patients who received at least 1 dose of the IMP. The SAF population was analyzed according to the actual treatment received and was used to present results on safety data.
Measure: Number; unit: number of adverse events
Groups:
- Total: The only investigational product administered in this study part, was Givinostat, therefore, all TEAEs were selected and reported upon.
Arm/Group | Total
Number analyzed (Participants) | 8
number of adverse events
  Total TEAE | 21
  mild TEAE | 17
  moderate TEAE | 4
  severe TEAE | 0

ADVERSE EVENTS:
Time Frame: Throughout the study and 10-14 days after the End of Study (follow-up visit), i.e. up to day 30-34, all TEAEs, considered related or not related to IMPs, were collected.
Description: End-of-study was defined as the last study procedure on Day 17 or at early discontinuation of subjects administered at least one dose of investigational product.
  Early termination procedures were performed as soon as possible after subject withdrawal, within 10-14 days after last participation of the subject in the study, whenever possible.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=8)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Bundle branch block right (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Migrane (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT05860114/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT05860114/SAP_001.pdf